CLINICAL TRIAL: NCT02270658
Title: Morbidity in Patients With Hypertension and Obstructive Sleep Apnea
Acronym: MORPHEOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Financiadora de Estudos e Projetos (Other); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Geraldo Lorenzi Filho, Principal Investigator, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3230/08/146
Record Dates: First submitted 2014-10-17; First posted 2014-10-21 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Hypertension; Sleep Apnea, Obstructive
Keywords: continuous positive airway pressure; hypertension; sleep apnea
MeSH Terms: conditions — Hypertension; Sleep Apnea, Obstructive; Sleep Apnea Syndromes | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Continuous positive airway pressure (Experimental): Continuous positive airway pressure therapy (CPAP)
  Interventions: Device: CPAP
- Nasal strips (Placebo Comparator): Nasal strips applied to the outside surface of the nose with adhesive.
  Interventions: Device: CPAP

INTERVENTIONS:
Device: CPAP
  Other Names: Continuous positive airway pressure

SUMMARY:
MORPHEOS is a multicenter, randomized, unblinded study, for patients diagnosed with uncontrolled hypertension and at least one antihypertensive medication. Those patients with significant sleep apnea wil be randomized to CPAP or nasal strips for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Systolic blood pressure ≥140 mm Hg or diastolic blood pressure ≥ 90 mm Hg
* Current treatment with at least 1 antihypertensive drug

Exclusion Criteria:

* Age <18 and >65 years
* BMI ≥ 40 kg/m2
* Heart failure, EF < 45%, acute myocardial infarction, stroke, significant valvular dysfunction
* Chronic renal failure (serum creatinine > 2 mg/dL)
* Use of cocaine, amphetamines, alcohol, illicit drugs
* Use of sympathomimetics (decongestants, appetite suppressants)
* Use of oral contraceptives and chronic use of NSAIDs
* Pregnancy
* Secondary causes of hypertension (other than sleep apnea)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Impact of OSA treatment with CPAP on office, 24-hour, and central blood pressure (co-primary endpoints). | 6 months

SECONDARY OUTCOMES:
Impact of OSA treatment with CPAP on target-organ damage | 6 months
Impact of OSA treatment with CPAP on vascular parameters (to be published as a sub-study) | 6 months
  Pulse wave velocity and carotid intima-media thickness
Impact of OSA treatment with CPAP on hypertensive retinopathy and optic nerve damage (to be published as a sub-study) | 6 months
Validation of portable sleep monitoring to diagnose OSA (to be published as a sub-study) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Geraldo Lorenzi, M.D. PhD, Principal Investigator — Fundação Zerbini - Instituto do Coração (InCor)
Locations (5):
- Brazil (5):
  - Pronto Socorro Cardiológico de Pernambuco (PROCAPE), Recife, Pernambuco
  - Hospital das Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto, Ribeirão Preto, São Paulo
  - Fundação Zerbini - Instituto do Coração (InCor), São Paulo, São Paulo
  - Hospital Universitário da Universidade de São Paulo (HU), São Paulo, São Paulo

REFERENCES:
- [Result] Cruz FCSG, Drager LF, Queiroz DBC, Souza GA, Pedrosa RP, Patriota TLGC, Dorea EL, Vieira MLC, Righi CG, Martinez D, Silva GAD, Silva GV, Pio-Abreu A, Lotufo PA, Benseaor IM, Bortolotto LA, Fuchs FD, Lorenzi-Filho G. The effect of continuous positive airway pressure on blood pressure in patients with obstructive sleep apnea and uncontrolled hypertension - Study design and challenges during the COVID-19 pandemic. Clinics (Sao Paulo). 2021 Sep 3;76:e2926. doi: 10.6061/clinics/2021/e2926. eCollection 2021. PMID 34495079
- [Derived] Lorenzi-Filho G, Cruz FCSG, Queiroz DBC, Vieira MLC, Pedrosa RP, Couto Patriota TLG, Righi CG, Martinez D, da Silva GA, Silva GV, Pio-Abreu A, Cabrini ML, Giampa SQC, Dorea EL, Lotufo PA, Bensenor IM, Bortolotto LA, Fuchs FD, Drager LF. Effects of Continuous Positive Airway Pressure on Central and Peripheral Blood Pressure in Patients with Uncontrolled Hypertension and Obstructive Sleep Apnea: The Randomized Controlled MORPHEOS Clinical Trial. Ann Am Thorac Soc. 2025 May;22(5):757-767. doi: 10.1513/AnnalsATS.202407-688OC. PMID 39879540